CLINICAL TRIAL: NCT01740518
Title: Randomized Controlled Trial of Low-volume PEG Plus Ascorbic Acid Versus Standard PEG Solution as Bowel Cleansing for Colonoscopy
Brief Title: Comparison of Low-volume PEG Plus Ascorbic Acid Versus Standard PEG Solution as Bowel Cleansing for Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dong Il Park, M.D, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Dong Il Park, M.D, Ph.D., associate professor, Kangbuk Samsung Hospital
Organization: Kangbuk Samsung Hospital (Other)
Other Study IDs: ASCPD
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Colonoscopy [E01.370.372.250.250.200]
MeSH Terms: interventions — Polyethylene Glycols; Ascorbic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PEG + ascorbic acid: Those who taken PEG 2L + ascorbic acid
  Interventions: Drug: polyethylene glycol, ascorbic acid
- PEG 4L: Those who taken PEG 4L alone

INTERVENTIONS:
Drug: polyethylene glycol, ascorbic acid — comparison of different solutions for bowel preparation
  Groups: PEG + ascorbic acid

SUMMARY:
The purpose of this study is to compare two regimens of low volume (2L) polyethylene glycol(PEG)plus ascorbic acid versus standard volume (4L) PEG alone for bowel preparation in out-patients

DETAILED DESCRIPTION:
Inadequate bowel preparation may lead to a longer colonoscopy, and to an inability to identify lesions. PEG can provide a rapid orthograde peroral approach to colonic lavage without producing significant fluid or electrolyte changes. Thus PEG is now commonly used for bowel preparation. However, large amounts and unsatisfactory taste of PEG solution are generally poorly tolerated. a new low volume PEG-based bowel cleansing agents became available at foreign countries. Although several studies reported the efficacy and improved compliance of these low volume PEG plus ascorbic acid solution for colonoscopy, but result in Korean patients was not-recognized.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients for colonoscopy

Exclusion Criteria:

* age under 19 years or over 80 years
* Intestinal obstruction
* Women of pregnant, breastfeeding, or at risk of becoming pregnant
* major psychiatric illness
* known allergy to PEG
* serious condition- severe cardiac, renal, or metabolic diseases
* past history of colon resection
* current acute exacerbation of chronic inflammatory bowel disease
* functional constipation defined by Rome III diagnostic criteria

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Out-patients for colonoscopy in university hospital
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of bowel preparation | one day (after colonoscopy)
  three segmental preparation scoring (0~4, Rt., mid, Lt.colon) total preparation grade:A,B,C,D (A or B was defined successful bowel cleansing) Influence of the intake of additional fluid in PEG+ascorbic acid

SECONDARY OUTCOMES:
Patient's compliance and acceptability | one day (after injestion of preparation solution)
  satisfaction (Visual Analogue Scale) amount of ingestion, frequency and amount of vomiting, tolerability, complication, taste

CONTACTS AND LOCATIONS:
Overall Officials: Dong Il Park, professor, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, Seoul, South Korea

REFERENCES:
- See also: Related Info — http://irb.kbsmc.co.kr